CLINICAL TRIAL: NCT03579602
Title: A Randomized, Blinded Study of Fluorescence Detection of Pediatric Primary Central Nervous System Tumors in Subjects Receiving Tozuleristide and Imaged With the Canvas System
Brief Title: Study of Tozuleristide and the Canvas Imaging System in Pediatric Subjects With CNS Tumors Undergoing Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Blaze Bioscience Inc. (Industry)
Collaborators: Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BB-006; PNOC012 (Other: Pacific Pediatric Neuro-Oncology Consortium)
Expanded Access: NCT04343274 (No longer available)
Record Dates: First submitted 2018-06-15; First posted 2018-07-06 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Central Nervous System Tumor
Keywords: Tumor Paint; tozuleristide; Canvas imaging system; BLZ-100; CNS tumor; brain cancer; pediatrics; fluorescence guided surgery
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — tozuleristide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:10 to 1 of 2 study arms. Subjects in arm 1 (~9% of subjects) will not receive tozuleristide but will undergo neurosurgery and imaging will be performed with the Canvas. Subjects in arm 2 (~91% of subjects) will receive tozuleristide and will undergo neurosurgery and imaging will be performed with the Canvas.
Who Masked: Outcomes Assessor
Masking Description: Central Pathology assessment and Central Radiology post-operative MRI assessment will be blinded to study arm and fluorescence data.
  Central Fluorescence assessment will be blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm 1 (no tozuleristide) (Active Comparator): Subjects randomized to Arm 1 (~9% of subjects) will not receive tozuleristide but will undergo standard of care neurosurgery and will have imaging performed with the Canvas System.
  Interventions: Device: Canvas System
- Arm 2 (tozuleristide treated) (Experimental): Subjects randomized to Arm 2 (~ 91% of subjects) will be administered tozuleristide at a dose of 15 mg/m^2 at least 1 hour and no more than 36 hours prior to surgery. They will undergo standard of care neurosurgery and will have imaging performed with the Canvas System.
  Interventions: Drug: tozuleristide; Device: Canvas System

INTERVENTIONS:
Drug: tozuleristide — Tozuleristide will be administered at least 1 hour and no more than 36 hours prior to planned surgical excision of their tumor.
  Other Names: BLZ-100; Tumor Paint
  Arms: Arm 2 (tozuleristide treated)
Device: Canvas System — All subjects enrolled in the study will have their tissue imaged with the Canvas System.
  Other Names: mSIRIS

SUMMARY:
Many types of cancer are primarily treated with surgery and patient survival is directly related to the extent to which the tumor is able to be removed. It is often difficult for surgeons to distinguish tumor tissue from normal tissue or to detect tumor cells that have spread from the original tumor site, resulting in incomplete removal of the tumor and reduced patient survival. In some sites, such as the brain, it is critical to avoid damage to normal tissue around the tumor to prevent adverse effects of surgery on function. Tozuleristide is a drug that is thought to attach to tumor tissue and then fluoresces (glows) when a special light from the Canvas is shined on it. It is hypothesized that tozuleristide, when imaged with the Canvas, will improve surgical outcomes by allowing surgeons to visualize the edges of the tumor or other ambiguous tissue in real-time as they operate. The purpose of this study is to evaluate how well tozuleristide imaged with Canvas work at helping to distinguish between tumor and normal tissue during surgery in pediatric primary central nervous system tumors.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent, or have it provided by their legally acceptable representative, will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

Surgical excision will occur at least 1 hour and no more than 36 hours after tozuleristide administration. Surgery will be performed by a neurosurgeon and the Canvas will be operated by a designated Imaging Operator. Fluorescence of tumor and ambiguous tissue during surgery will be assessed and scored. Biopsy samples of these tumor and ambiguous tissues will be collected for pathology analysis.

All subjects will be monitored for safety during their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be >1 month and ≤30 years of age at the time of study enrollment
2. Subjects must have MRI obtained within 30 days of study enrollment documenting a measurable lesion consistent with a pediatric primary CNS tumor for which maximal safe resection is indicated
3. Adequate renal function
4. Adequate liver function
5. Prior therapy: Subjects with prior therapy are eligible provided they have recovered from any acute toxic effects of prior therapy and have sufficient time interval prior to enrollment:

   1. Radiation therapy: subjects may not have had radiation therapy to the area of tumor planned to be resected within 28 days of study enrollment
   2. Chemotherapy: at least 14 days from any myelosuppressive chemotherapy (28 days if prior nitrosourea) and if prior chemotherapy, must have an absolute neutrophil count recovery of ≥ 1000/mm3 following count nadir
   3. Biologic: at least 7 days from any anti-neoplastic biologic agent (at least 3 half-lives since last administration of monoclonal antibodies)
   4. Immunotherapy: at least 42 days after completion of any cellular immunotherapy, such as CAR-T cell therapy
   5. Prior surgery for CNS tumors is allowed
   6. Prior tozuleristide: at least 1 week after prior dose of tozuleristide if previously treated
6. Written informed consent must be obtained from the subject or parent or legal guardian prior to the conduct of study activities. Routine clinical tests, e.g., MRI, clinical laboratory studies, may be used for screening requirements. Assent, when appropriate, will be obtained according to institutional guidelines.
7. The risks of treatment with tozuleristide during pregnancy have not been evaluated. Female subjects of child-bearing potential must agree not to attempt to become pregnant or undergo in vitro fertilization and, if participating in sexual activity that could lead to pregnancy, must use 2 reliable methods of contraception simultaneously for 30 days after surgery. Male subjects must agree not to attempt to father a child and, if participating in sexual activity that could lead to pregnancy, must use 2 reliable methods of contraception simultaneously for 30 days after surgery if their partner is of child-bearing potential.

Exclusion Criteria:

1. Pregnancy and contraception: Subjects who are pregnant or breast-feeding or planning to conceive a child within 30 days are not eligible. Males and females of childbearing potential must agree to use 2 effective forms of contraception from the time of enrollment until 30 days post-surgery
2. Subjects with on-going serious medical conditions (poorly controlled asthma, diabetes, heart disease) such that participation in the study could put the subject at increased risk of worsening their condition
3. Subjects planned to undergo only a diagnostic biopsy procedure, without intent to resect tissue for therapeutic purposes (e.g., stereotactic pontine biopsy)
4. Subjects who in the opinion of the investigator are not willing or able to comply with randomization procedures or other study-required study procedures and observations. Subjects previously enrolled and randomized to Arm 1 (control) are not eligible for re-enrollment unless a second surgery is required by standard of care.

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Leary, MD, Principal Investigator — Seattle Children's Hospital
Locations (9):
- United States (9):
  - Chlidren's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Florida Shands Hospital, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Minnesota, Saint Paul, Minnesota
  - Washington University St. Louis Children's Hospital, St Louis, Missouri
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 118 subjects were enrolled from 9 academic sites
Period: Overall Study
Arm/Group | Arm 1 (no Tozuleristide) | Arm 2 (Tozuleristide Treated)
Started | 11 | 107
Subjects Who Received Tozuleristide Retreatment | 2 | 2
Completed | 11 | 104
Not Completed | 0 | 3
Not completed — Subject unable to receive study drug | 0 | 2
Not completed — Subject did not complete all study visits as planned | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study's safety analysis population is used for these baseline data. The safety analysis population consists of all subjects who receive any amount of tozuleristide or receive neurosurgery prior to any re-treatment. There were two subjects from Arm 2 who were not dosed with tozuleristide which is the reason the Overall Number of Baseline Participants (n=116) is two less than the # of patients entered into the Total Started in Participant Flow: (n=118).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (no Tozuleristide) | Arm 2 (Tozuleristide Treated) | Total
Number analyzed (Participants) | 11 | 105 | 116
Age, Continuous [Mean (Full Range); unit: years] | 7.749 [3.07 to 12.90] | 9.445 [0.31 to 27.12] | 9.284 [0.31 to 27.12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 40 | 45
  Male | 6 | 65 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 10 | 10
  Ethnicity: Not Hispanic or Latino | 7 | 72 | 79
  Ethnicity: Unknown or Not Reported | 4 | 23 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 1 | 12 | 13
  White | 8 | 71 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 10 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 105 | 116
Weight [Mean (Full Range); unit: kg] | 27.09 [11.9 to 35.9] | 37.14 [6.2 to 126.5] | 36.19 [6.2 to 126.5]
Height [Mean (Full Range); unit: cm] | 121.72 [78.7 to 148.0] | 130.46 [61.0 to 185.8] | 129.63 [61.0 to 185.8]
BSA [Mean (Full Range); unit: m sq] | 0.9534 [0.510 to 1.215] | 1.1351 [0.329 to 2.458] | 1.1178 [0.329 to 2.458]
Karnofsky Performance Status Score [Count of Participants; unit: Participants] — 100 Normal, no complaints, no evidence of disease; 90 Able to carry on normal activity, minor signs of symptoms of disease; 80 Normal activity with effort, some signs or symptoms of disease; 70 Cares for self, unable to carry on normal activity or do active work; 60 Requires occasional assistance, but is able to care for most of his/her needs; 50 Requires considerable assistance and frequent medical care; 40 Disabled, requires special care and assistance Population: Enrolled participants were assessed according to either the Karnofsky Performance Status Score OR the Lansky Performance Status Score (not both). 28 out of the 116 participants enrolled into the study completed the Karnofsky Performance Status Score and 88 out of the 116 participants enrolled into the study completed the Lanksy Performance Status Score. (28 Lansky Assessments + 88 Karnofsky Assessments = 116 assessments [1 for each participant enrolled into the study])
  Participants
    100: number analyzed (Participants) | 2 | 26 | 28
    100 | 0 | 12 | 12
    90: number analyzed (Participants) | 2 | 26 | 28
    90 | 2 | 4 | 6
    80: number analyzed (Participants) | 2 | 26 | 28
    80 | 0 | 6 | 6
    70: number analyzed (Participants) | 2 | 26 | 28
    70 | 0 | 1 | 1
    50: number analyzed (Participants) | 2 | 26 | 28
    50 | 0 | 2 | 2
    40: number analyzed (Participants) | 2 | 26 | 28
    40 | 0 | 1 | 1
Lansky Performance Status Score [Count of Participants; unit: Participants] — Uses parent description of child's activity to assess ability and response to treatment. 100 Fully active, normal; 90 Minor restrictions in physically strenuous activity; 80 Actives, but tires more quickly; 70 Both greater restriction of and less time spent in play activity; 60 Up and around, but minimal active play; keeps busy with quieter activities; 50 Gets dressed, but lies around much of the day; no active play, able to participate in all quiet play and activities; 40 Mostly in bed; participates in quiet activities; 30 Needs considerable assistance for quiet activity Population: Enrolled participants were assessed according to either the Karnofsky Performance Status Score OR the Lansky Performance Status Score (not both). 28 out of the 116 participants enrolled into the study completed the Karnofsky Performance Status Score and 88 out of the 116 participants enrolled into the study completed the Lanksy Performance Status Score. (28 Lansky Assessments + 88 Karnofsky Assessments = 116 assessments [1 for each participant enrolled into the study])
  Participants
    100: number analyzed (Participants) | 9 | 79 | 88
    100 | 5 | 38 | 43
    90: number analyzed (Participants) | 9 | 79 | 88
    90 | 1 | 25 | 26
    80: number analyzed (Participants) | 9 | 79 | 88
    80 | 2 | 9 | 11
    70: number analyzed (Participants) | 9 | 79 | 88
    70 | 1 | 6 | 7
    30: number analyzed (Participants) | 9 | 79 | 88
    30 | 0 | 1 | 1
Received Prior CNS Cancer Surgery [Count of Participants; unit: Participants]
  Yes | 3 | 38 | 41
  No | 8 | 67 | 75
Received Prior CNS Cancer Systemic Therapy, [Count of Participants; unit: Participants]
  Yes | 1 | 22 | 23
  No | 10 | 83 | 93
Received Prior CNS Cancer Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 1 | 14 | 15
  No | 10 | 91 | 101
Recurrent or Progressive Disease for Current Tumor [Count of Participants; unit: Participants]
  Yes | 3 | 33 | 36
  No | 8 | 72 | 80
Evidence of Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 0 | 10 | 10
  No | 11 | 91 | 102
  Unknown | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Tozuleristide Fluorescence to Detect Tumor in Equivocal (Ambiguous) Tissue During Surgery When Imaged With the Canvas System
Description: Sensitivity and specificity of tozuleristide imaged with the Canvas system to fluorescently identify tumor in equivocal tissue will be evaluated based on central pathology consensus assessment of tumor and by imaging operator fluorescence assessment. These measures will be compared to the sensitivity and specificity of surgical designation of tumor (more likely tumor or less likely tumor) under white light. Sensitivity reflects the probability that tumor tissue evaluated is fluorescent. Specificity reflects the probability that normal tissue evaluated is not fluorescent. Equivocal tissues are those that the surgeon considers abnormal but ambiguous as tumor vs. not tumor under normal (white light) conditions.
Time Frame: During surgery (which occurs at least 1 hour post tozuleristide administration)
Population: (Group 2) Subjects who receive tozuleristide, have at least one fluorescence-positive study tissue specimens of any type (primary, equivocal, and other) based on imaging operator fluorescence assessment, and the subject's central pathology consensus diagnosis is tumor, ambiguous, or not definitive.
Measure: Number (95% Confidence Interval); unit: % of equivocal tissue biopsies
Units Other Than Participants: Equivocal Tissue Biopsies
Groups:
- Group 2: Group 2 (Arm 2 Fluorescent): subjects who receive tozuleristide, have at least one fluorescence-positive study tissue specimens of any type (primary, equivocal and other) based on imaging operator fluorescence assessment, and the subject's central pathology consensus diagnosis is tumor, ambiguous, or not definitive
Arm/Group | Group 2
Number analyzed (Participants) | 61
Number analyzed (Equivocal Tissue Biopsies) | 156
% of equivocal tissue biopsies
  Sensitivity of Tozuleristide Fluorescence for equivocal tissue biopsies in Group 2 | 79.8 [70.2 to 90.9]
  Specificity of Tozuleristide Fluorescence for equivocal tissue biopsies in Group 2 | 34.7 [22.5 to 53.6]

2. Primary Outcome: Ratio of Tozuleristide Sensitivity Compared to Surgeon Sensitivity
Description: Tozuleristide sensitivity as assessed by imaging operator fluorescence assessment compared to sensitivity of surgeon designation of tumor under white light in equivocal tissue biopsies. Sensitivity reflects the probability that tumor tissue evaluated is fluorescent. Equivocal tissues are those that the surgeon considers abnormal but ambiguous as tumor vs. not tumor under normal (white light) conditions.
Time Frame: During surgery (which occurs at least 1 hour post tozuleristide administration)
Population: Subjects who receive tozuleristide, have at least one fluorescence-positive study tissue specimens of any type (primary, equivocal, and other) based on imaging operator fluorescence assessment, and the subject's central pathology consensus diagnosis is tumor, ambiguous, or not definitive.
Measure: Number (95% Confidence Interval); unit: Ratio of sensitivity
Units Other Than Participants: Equivocal Tissue Biopsies
Arm/Group | Group 2
Number analyzed (Participants) | 61
Number analyzed (Equivocal Tissue Biopsies) | 156
Ratio of sensitivity | 1.099 [0.929 to 1.300]

3. Primary Outcome: Ratio of Tozuleristide Specificity Compared to Surgeon Specificity
Description: Tozuleristide specificity as assessed by imaging operator fluorescence assessment compared to specificity of surgeon designation of tumor under white light in equivocal tissue biopsies. Specificity reflects the probability that normal tissue evaluated is not fluorescent. Equivocal tissues are those that the surgeon considers abnormal but ambiguous as tumor vs. not tumor under normal (white light) conditions.
Time Frame: During surgery (which occurs at least 1 hour post tozuleristide administration)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Ratio of specificity
Units Other Than Participants: Equivocal Tissue Biopsies
Arm/Group | Group 2
Number analyzed (Participants) | 61
Number analyzed (Equivocal Tissue Biopsies) | 156
Ratio of specificity | 0.614 [0.348 to 1.083]

ADVERSE EVENTS:
Time Frame: From randomization through three months following surgery, or until start of other tumor-directed therapy, whichever is earlier, up to 3 months. Average time on study was approximately 9 weeks.
Description: Serious Adverse Events (AEs) includes all Serious AEs reported, none assessed related to tozuleristide by the investigator. Other AEs includes all treatment-emergent AEs reported in =>5% of subjects on Arm 1 (no tozuleristide) or Arm 2 (tozuleristide treated). Only the following 5 TEAEs were assessed related to tozuleristide by the investigator, occurring in 1 subject each (1/105 Arm 2 subjects, 0.95%): injection site joint pain, vomiting, proteinuria, hypoalbuminemia, maculopapular rash.
Arm/Group | Arm 1 (no Tozuleristide) | Arm 2 (Tozuleristide Treated)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/105
Serious Adverse Events (participants affected / at risk) | 4/11 | 28/105
Other Adverse Events (participants affected / at risk) | 11/11 | 105/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (no Tozuleristide) (N=11) | Arm 2 (Tozuleristide Treated) (N=105)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Depressed Level of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Facial Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Posterior fossa syndrome (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (no Tozuleristide) (N=11) | Arm 2 (Tozuleristide Treated) (N=105)
Constipation (Gastrointestinal disorders) | 4 | 38
Nausea (Gastrointestinal disorders) | 4 | 34
Vomiting (Gastrointestinal disorders) | 4 | 31
Dysphagia (Gastrointestinal disorders) | 0 | 6
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Glossitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 24
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 23
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 16
Decreased appetite (Metabolism and nutrition disorders) | 2 | 12
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 7
Alkalosis (Metabolism and nutrition disorders) | 2 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 7 | 52
Incision site pain (Injury, poisoning and procedural complications) | 2 | 9
Pseudomeningocele (Injury, poisoning and procedural complications) | 2 | 5
Incision site oedema (Injury, poisoning and procedural complications) | 2 | 3
Wound complication (Injury, poisoning and procedural complications) | 1 | 2
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 1
Incision site pruritus (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 61
Headache (Nervous system disorders) | 3 | 28
Ataxia (Nervous system disorders) | 3 | 10
Dizziness (Nervous system disorders) | 1 | 10
Dysarthria (Nervous system disorders) | 1 | 10
Hemiparesis (Nervous system disorders) | 1 | 8
Hydrocephalus (Nervous system disorders) | 1 | 6
Lethargy (Nervous system disorders) | 2 | 6
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 4
VIth nerve disorder (Nervous system disorders) | 1 | 3
Seizure (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 1 | 1
Basal ganglia stroke (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 31
Alanine aminotransferase increased (Investigations) | 1 | 17
Weight increased (Investigations) | 1 | 10
Blood bicarbonate decreased (Investigations) | 1 | 9
Weight decreased (Investigations) | 2 | 6
White blood cell count decreased (Investigations) | 1 | 4
Breath sounds abnormal (Investigations) | 1 | 0
Fatigue (General disorders) | 3 | 21
Pyrexia (General disorders) | 3 | 18
Face oedema (General disorders) | 2 | 6
Pain (General disorders) | 1 | 5
Asthenia (General disorders) | 2 | 3
Generalised oedema (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 11
Agitation (Psychiatric disorders) | 2 | 9
Anxiety (Psychiatric disorders) | 1 | 8
Insomnia (Psychiatric disorders) | 1 | 5
Confusional state (Psychiatric disorders) | 1 | 3
Delirium (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 1 | 3
Restlessness (Psychiatric disorders) | 1 | 3
Delusion (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 2 | 0
Periorbital oedema (Eye disorders) | 1 | 12
Vision blurred (Eye disorders) | 1 | 8
Diplopia (Eye disorders) | 1 | 4
Eye pain (Eye disorders) | 1 | 2
Anisocoria (Eye disorders) | 1 | 1
Eyelid ptosis (Eye disorders) | 1 | 1
Strabismus (Eye disorders) | 1 | 1
Lagophthalmos (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 19
Sinus bradycardia (Cardiac disorders) | 1 | 8
Sinus tachycardia (Cardiac disorders) | 0 | 8
Bradycardia (Cardiac disorders) | 1 | 4
Tachycardia (Cardiac disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 7
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Candida infection (Infections and infestations) | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03579602/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT03579602/SAP_002.pdf